CLINICAL TRIAL: NCT00528957
Title: A Phase III, Randomized, Open-Label Study Comparing the Safety and Efficacy of Switching Stavudine or Zidovudine to Tenofovir Disoproxil Fumarate Versus Continuing Stavudine or Zidovudine in Virologically Suppressed HIV-Infected Children Taking Highly Active Antiretroviral Therapy
Brief Title: Safety and Efficacy of Switching From Stavudine or Zidovudine to Tenofovir DF in HIV-1 Infected Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-104-0352; 2007-003418-32 (EudraCT Number)
Record Dates: First submitted 2007-01-03; First posted 2007-09-14 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
Keywords: Phase 3; Randomized, Open-Label; Treatment-Experienced; Highly Active Antiretroviral Therapy; HIV; Tenofovir DF; Pediatrics
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Zidovudine; Stavudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenofovir DF (Experimental)
  Interventions: Drug: Tenofovir DF
- stavudine or zidovudine (Active Comparator)
  Interventions: Drug: Zidovudine; Drug: Stavudine

INTERVENTIONS:
Drug: Tenofovir DF — Tenofovir DF (oral powder or tablet): 300-mg tablets for participants > 37 kg; 8-mg/kg oral powder (up to 300 mg) for participants ≤ 37 kg. During the extension phase, participants whose weight increases to > 37 kg may be switched from the oral powder to the tenofovir DF tablet.
  Other Names: Viread®
  Arms: Tenofovir DF
Drug: Zidovudine — Zidovudine as prescribed by the investigator prior to study entry (pediatric participants < 30 kg: 1 mg/kg/dose given every 12 hours; pediatric participants ≥ 30 kg: 30 mg twice daily).
  Arms: stavudine or zidovudine
Drug: Stavudine — Stavudine as prescribed by the investigator prior to study entry (pediatric participants 6 weeks to 12 years of age: 160 mg/m^2 every 8 hours; pediatric participants > 12 years of age: 300 mg twice daily).
  Arms: stavudine or zidovudine

SUMMARY:
The primary objective of this study is to assess the efficacy of switching to tenofovir disoproxil fumarate (TDF) compared to continuing stavudine or zidovudine in maintaining virologic suppression in HIV-1 infected children.

ELIGIBILITY:
Major Inclusion Criteria:

* Documented laboratory diagnosis of HIV-1 infection
* Plasma HIV-1 RNA < 400 copies/mL
* Currently on a stable stavudine or zidovudine -containing antiretroviral therapy regimen for at least 12 weeks
* Naive to tenofovir DF

Key Inclusion Criteria for the First 96-Week Extension

* Completed 48 weeks of treatment in Arm 1 or Arm 2 of the study
* <18 years of age (at the start of the extension)
* Participants initially randomized to Arm 2 will be given the option to replace stavudine or zidovudine with tenofovir DF in the 96-week extension at the investigator's discretion, if the investigator determines that tenofovir DF is safe and beneficial for the participant.

Key Inclusion Criteria for the Second and Third 96-Week Extension and Fourth Open-Ended Extension

* Completed of treatment with study drug in the first extension phase
* <18 years of age at the start of the extension. This inclusion criterion is not applicable in those regions where tenofovir DF is not commercially available for treatment of HIV-1 infection in adults.

Key Exclusion Criteria:

* Participants receiving ongoing therapy with any of the following
* Nephrotoxic agents
* Systemic chemotherapeutic agents
* Systemic corticosteroids
* Interleukin 2 (IL 2) and other immunomodulating agents
* Investigational agents
* Pregnant or lactating participants
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic therapy within 15 days prior to screening
* Prior history of significant renal disease (ie, nephrotic syndrome, renal dysgenesis, polycystic kidney disease, congenital nephrosis)
* Prior history of significant bone disease (ie, osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochondroses, multiple bone fractures)

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2006-12-28 (Actual); Primary Completion 2009-04-06 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- United States (6):
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - University California Los Angeles, School of Medicine, Pediatric, Infectious Diseases, Los Angeles, California
  - Children's Diagnostic and Treatment Center, Inc, Fort Lauderdale, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Hospital del Nino, Panama City, Panama
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Imperial College London, Paediatrics Infectious Diseases, London

REFERENCES:
- [Derived] Saez-Llorens X, Castano E, Rathore M, Church J, Deville J, Gaur A, Estripeaut D, White K, Arterburn S, Enejosa JV, Cheng AK, Chuck SL, Rhee MS. A randomized, open-label study of the safety and efficacy of switching stavudine or zidovudine to tenofovir disoproxil fumarate in HIV-1-infected children with virologic suppression. Pediatr Infect Dis J. 2015 Apr;34(4):376-82. doi: 10.1097/INF.0000000000000289. PMID 25760565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Panama, and the United Kingdom. The first participant was screened on 28 December 2006. The last study visit occurred on 16 August 2017.
Pre-assignment Details: 127 participants were screened.
Groups:
- Tenofovir DF: Participants in this group received tenofovir disoproxil fumarate (TDF) during the randomized phase (48 weeks) and continued to receive TDF during the extension phase(s).
- Stavudine or Zidovudine: Participants in this group received stavudine or zidovudine during the randomized phase (48 weeks) and then received TDF during the extension phase(s).
Period: Randomized Phase (Baseline to Week 48)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Started | 48 | 49
Completed | 44 | 48
Not Completed | 4 | 1
Not completed — Withdrew Consent | 2 | 1
Not completed — Safety, Tolerability, or Efficacy Reason | 2 | 0
Period: First Extension (Week 48 to Week 144)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Started | 38 (Six participants completed the 48-week randomized phase and did not enroll in the first extension.) | 41 (Seven participants completed the 48-week randomized phase and did not enroll in the first extension.)
Completed | 35 | 40
Not Completed | 3 | 1
Not completed — Investigator's Discretion | 2 | 0
Not completed — Safety, Tolerability, or Efficacy Reason | 1 | 0
Not completed — Withdrew Consent | 0 | 1
Period: Second Extension (Week 144 to Week 240)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Started | 34 (One participant completed the first extension and did not enroll in the second extension.) | 40
Completed | 27 | 37
Not Completed | 7 | 3
Not completed — Safety, Tolerability, or Efficacy Reason | 4 | 3
Not completed — Investigator's Discretion | 3 | 0
Period: Third Extension (Week 240 to Week 336)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Started | 27 | 37
Completed | 21 | 27
Not Completed | 6 | 10
Not completed — Safety, Tolerability, or Efficacy Reason | 5 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — = 18 yr old & TDF approved in adults | 1 | 1
Not completed — Investigator's Discretion | 0 | 1
Not completed — Withdrew Consent | 0 | 1
Period: Long-Term Extension (Week 336 and On)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Started | 19 (Two participants completed the third extension and did not enroll in the long-term extension.) | 25 (Two participants completed the third extension and did not enroll in the long-term extension.)
Completed | 9 | 8
Not Completed | 10 | 17
Not completed — Rolled Over to Study GS-US-311-1269 | 4 | 10
Not completed — Safety, Tolerability, or Efficacy Reason | 3 | 5
Not completed — Withdrew Consent | 2 | 1
Not completed — Investigator's Discretion | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized and Treated Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- Tenofovir DF: Participants in this group received TDF during the randomized phase (48 weeks) and continued to receive TDF during the extension phase(s).
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (3.3) | 7 (2.6) | 7 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 20 | 47
  Male | 21 | 29 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 42 | 77
  Not Hispanic or Latino | 13 | 7 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 3 | 6 | 9
  Mestizo | 28 | 37 | 65
  Native Indian (Kuna) | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 9 | 22
  Panama | 33 | 39 | 72
  United Kingdom | 2 | 1 | 3
Height [Mean (Standard Deviation); unit: cm] | 118 (19.8) | 119 (16.7) | 119 (18.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 17.59 (3.680) | 16.59 (1.762) | 17.08 (2.905)
Weight [Mean (Standard Deviation); unit: kilograms] | 25.9 (12.03) | 24.1 (7.77) | 25.0 (10.09)
Plasma HIV-1 RNA [Count of Participants; unit: Participants]
  < 50 copies/mL | 36 | 41 | 77
  50 to < 400 copies/mL | 11 | 6 | 17
  400 to < 1000 copies/mL | 1 | 1 | 2
  ≥ 1000 copies/mL | 0 | 1 | 1
CD4 Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 1190 (541.7) | 1144 (388.4) | 1167 (468.6)
CD4 Percentage [Mean (Standard Deviation); unit: percentage] | 33.9 (7.44) | 33.0 (6.82) | 33.5 (7.11)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 48
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 48 weeks of exposure to randomized study drug.
Time Frame: 48 weeks
Population: Intent-to-treat, Missing = Failure
Measure: Number; unit: percentage of participants
Groups:
- Tenofovir DF: Participants in this group received TDF during the randomized phase (48 weeks)
- Stavudine or Zidovudine: Participants in this group received stavudine or zidovudine during the randomized phase (48 weeks)
- All TDF: All participants who received tenofovir DF in the randomized and/or extension phases
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | All TDF
Number analyzed (Participants) | 48 | 49 | 89
percentage of participants | 83.3 [69.8 to 92.5] | 91.8 [80.4 to 97.7] | 85.4 [76.3 to 92.0]
Statistical Analysis 1: Comparison: Tenofovir DF vs Stavudine or Zidovudine; The statistical hypotheses for the primary endpoint was as follows: * Null Hypothesis: tenofovir DF group is more than 15% worse than the stavudine or zidovudine group with respect to the proportion of participants maintaining HIV-1 RNA concentrations < 400 copies/mL at Week 48. * Alternate Hypothesis: tenofovir DF group is no more than 15% worse than the stavudine or zidovudine group with respect to the proportion of participants maintaining HIV-1 RNA < 400 copies/mL at Week 48; Test type: Non-Inferiority or Equivalence — In the randomized phase, it was assumed that the respective proportions of participants maintaining HIV-1 RNA < 400 copies/mL was 92% for participants switching to tenofovir DF and 90% for participants continuing stavudine or zidovudine, as estimated from previous GSI studies. The equivalence limit was set at -15% for the lower boundary of a two-sided 95% confidence interval (CI) on the difference in proportions of participants maintaining HIV-1 RNA < 400 copies/mL at Week 48; Normal approximation; The difference between the two proportions and its CI were based on normal approximation methods; Difference in percentages between groups = -8.5, 95% CI 2-sided [-21.5 to 4.5] — Difference is for tenofovir DF minus stavudine or zidovudine (randomized phase)

2. Secondary Outcome: Virologic Success at 48 Weeks (HIV-1 RNA Cutoff at 400 Copies/mL, Snapshot)
Description: This is the percentage of participants with virologic success after 48 weeks of exposure to randomized study drug. The percentage of participants achieving HIV-1 RNA < 400 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: 48 weeks
Population: Intent-to-treat (ITT) Analysis Set; only includes participants < 12 years of age at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Number analyzed (Participants) | 44 | 48
percentage of participants | 88.6 | 89.6
Statistical Analysis 1: Comparison: Tenofovir DF vs Stavudine or Zidovudine; Test type: Non-Inferiority — In the randomized phase, it was assumed that the respective proportions of participants maintaining HIV-1 RNA < 400 copies/mL was 92% for subjects switching to tenofovir DF and 90% for subjects continuing stavudine or zidovudine, as estimated from previous GSI studies. The equivalence limit was set at -15% for the lower boundary of a two-sided 95% confidence interval (CI) on the difference in proportions of participants maintaining HIV-1 RNA < 400 copies/mL at Week 48; Difference in percentages between groups = -0.9, 95% CI 2-sided [-13.7 to 11.8] — The difference between the two proportions and its CI were based on normal approximation methods

3. Secondary Outcome: Virologic Success at 48 Weeks (HIV-1 RNA Cutoff at 50 Copies/mL, Snapshot)
Description: This is the percentage of participants with virologic success after 48 weeks of exposure to randomized study drug. The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: 48 weeks
Population: Intent-to-treat (ITT) Analysis Set; only includes participants < 12 years of age at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Stavudine or Zidovudine
Number analyzed (Participants) | 44 | 48
percentage of participants | 75.0 | 81.3

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 96
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 96 weeks of exposure to TDF.
Time Frame: 96 weeks
Population: Intent-to-treat, Missing = Failure. Participants who had not reached the upper limit of the analysis window (date varies depending on analysis time frame) were excluded.
Measure: Number; unit: percentage of participants
Groups:
- (Stavudine or Zidovudine)/TDF: Participants in this group received stavudine or zidovudine during the randomized phase (48 weeks) and then received TDF during the extension phase(s)
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 38 | 41 | 79
percentage of participants | 81.6 | 85.4 | 83.5

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 144
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 144 weeks of exposure to TDF.
Time Frame: 144 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- All TDF: All participants who received tenofovir DF in the randomized and/or extension phases (All TDF group)
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 38 | 40 | 78
percentage of participants | 73.7 | 87.5 | 80.8

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 192 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 192 weeks of exposure to TDF.
Time Frame: 192 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- All TDF: All participants who received TDF in the randomized and/or extension phases (All TDF group)
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 34 | 40 | 74
percentage of participants | 70.6 | 82.5 | 77.0

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 240 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 240 weeks of exposure to TDF.
Time Frame: 240 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 34 | 37 | 71
percentage of participants | 70.6 | 75.7 | 73.2

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 288 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 288 weeks of exposure to TDF.
Time Frame: 288 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 27 | 37 | 64
percentage of participants | 81.5 | 67.6 | 73.4

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 336 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 336 weeks of exposure to TDF.
Time Frame: 336 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 22 | 21 | 43
percentage of participants | 90.9 | 100.0 | 95.3

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 384 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 384 weeks of exposure to TDF.
Time Frame: 384 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 17 | 9 | 26
percentage of participants | 100.0 | 100.0 | 100.0

11. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 432 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 432 weeks of exposure to TDF.
Time Frame: 432 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 13 | 7 | 20
percentage of participants | 100.0 | 85.7 | 95.0

12. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 480 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 480 weeks of exposure to TDF.
Time Frame: 480 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 9 | 2 | 11
percentage of participants | 88.9 | 100.0 | 90.9

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at 528 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 400 copies/mL after 528 weeks of exposure to TDF.
Time Frame: 528 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 6 | 0 | 6
percentage of participants | 100.0 |  | 100.0

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 48 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 48 weeks of exposure to randomized study drug.
Time Frame: 48 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | All TDF
Number analyzed (Participants) | 48 | 49 | 89
percentage of participants | 70.8 | 85.7 | 68.5

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 96 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 96 weeks of exposure to TDF.
Time Frame: 96 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 38 | 41 | 79
percentage of participants | 76.3 | 68.3 | 72.2

16. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 144 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 144 weeks of exposure to TDF.
Time Frame: 144 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 38 | 40 | 78
percentage of participants | 63.2 | 75.0 | 69.2

17. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 192 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 192 weeks of exposure to TDF.
Time Frame: 192 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 34 | 40 | 74
percentage of participants | 67.6 | 75.0 | 71.6

18. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 240 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 240 weeks of exposure to TDF.
Time Frame: 240 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 34 | 37 | 71
percentage of participants | 70.6 | 73.0 | 71.8

19. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 288 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 288 weeks of exposure to TDF.
Time Frame: 288 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 27 | 37 | 64
percentage of participants | 81.5 | 62.2 | 70.3

20. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 336 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 336 weeks of exposure to TDF.
Time Frame: 336 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 22 | 21 | 43
percentage of participants | 86.4 | 90.5 | 88.4

21. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 384 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 384 weeks of exposure to TDF.
Time Frame: 384 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 17 | 9 | 26
percentage of participants | 88.2 | 100.0 | 92.3

22. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 432 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 432 weeks of exposure to TDF.
Time Frame: 432 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 13 | 7 | 20
percentage of participants | 100.0 | 71.4 | 90.0

23. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 480 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 480 weeks of exposure to TDF.
Time Frame: 480 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 9 | 2 | 11
percentage of participants | 77.8 | 50.0 | 72.7

24. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at 528 Weeks
Description: This is the percentage of participants with HIV-1 RNA < 50 copies/mL after 528 weeks of exposure to TDF.
Time Frame: 528 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 6 | 0 | 6
percentage of participants | 100.0 |  | 100.0

25. Secondary Outcome: Change From Baseline in CD4 Percentage at 48 Weeks
Description: This is the change from baseline in CD4 percentage after 48 weeks of exposure to randomized study drug.
Time Frame: Baseline and 48 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | All TDF
Number analyzed (Participants) | 46 | 48 | 86
percentage | 0.3 (4.49) | 1.1 (4.73) | 0.6 (3.85)

26. Secondary Outcome: Change From Baseline in CD4 Percentage at 96 Weeks
Description: This is the change from baseline in CD4 percentage after 96 weeks of exposure to TDF.
Time Frame: Baseline and 96 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 37 | 38 | 75
percentage | 1.3 (4.08) | -0.1 (3.60) | 0.6 (3.88)

27. Secondary Outcome: Change From Baseline in CD4 Percentage at 144 Weeks
Description: This is the change from baseline in CD4 percentage after 144 weeks of exposure to TDF.
Time Frame: Baseline and 144 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 33 | 38 | 71
percentage | 0.8 (5.61) | -0.1 (3.83) | 0.3 (4.73)

28. Secondary Outcome: Change From Baseline in CD4 Percentage at 192 Weeks
Description: This is the change from baseline in CD4 percentage after 192 weeks of exposure to TDF.
Time Frame: Baseline and 192 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 29 | 37 | 66
percentage | 1.1 (5.57) | 0.6 (3.69) | 0.8 (4.58)

29. Secondary Outcome: Change From Baseline in CD4 Percentage at 240 Weeks
Description: This is the change from baseline in CD4 percentage after 240 weeks of exposure to TDF.
Time Frame: Baseline and 240 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 28 | 32 | 60
percentage | 1.3 (5.98) | -0.9 (4.13) | 0.1 (5.16)

30. Secondary Outcome: Change From Baseline in CD4 Percentage at 288 Weeks
Description: This is the change from baseline in CD4 percentage after 288 weeks of exposure to TDF.
Time Frame: Baseline and 288 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 26 | 26 | 52
percentage | 2.0 (6.30) | 0.5 (4.77) | 1.3 (5.58)

31. Secondary Outcome: Change From Baseline in CD4 Percentage at 336 Weeks
Description: This is the change from baseline in CD4 percentage after 336 weeks of exposure to TDF.
Time Frame: Baseline and 336 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 23 | 22 | 45
percentage | 2.0 (7.19) | 0.8 (4.01) | 1.4 (5.82)

32. Secondary Outcome: Change From Baseline in CD4 Percentage at 384 Weeks
Description: This is the change from baseline in CD4 percentage after 384 weeks of exposure to TDF.
Time Frame: Baseline and 384 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 19 | 10 | 29
percentage | 0.5 (7.80) | 1.6 (1.90) | 0.9 (6.37)

33. Secondary Outcome: Change From Baseline in CD4 Percentage at 432 Weeks
Description: This is the change from baseline in CD4 percentage after 432 weeks of exposure to TDF.
Time Frame: Baseline and 432 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 14 | 7 | 21
percentage | 0.3 (6.41) | 2.9 (3.53) | 1.1 (5.66)

34. Secondary Outcome: Change From Baseline in CD4 Percentage at 480 Weeks
Description: This is the change from baseline in CD4 percentage after 480 weeks of exposure to TDF.
Time Frame: Baseline and 480 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 10 | 3 | 13
percentage | 2.3 (7.15) | 5.0 (10.00) | 2.9 (7.51)

35. Secondary Outcome: Change From Baseline in CD4 Percentage at 528 Weeks
Description: This is the change from baseline in CD4 percentage after 528 weeks of exposure to TDF.
Time Frame: Baseline and 528 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 6 | 0 | 6
percentage | 4.5 (3.89) |  | 4.5 (3.89)

36. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 48 Weeks
Description: This is the change from baseline in CD4 cell count after 48 weeks of exposure to randomized study drug.
Time Frame: Baseline and 48 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | All TDF
Number analyzed (Participants) | 46 | 48 | 86
cells/mm^3 | -97 (416.4) | -11 (280.2) | 2 (385.9)

37. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 96 Weeks
Description: This is the change from baseline in CD4 cell count after 96 weeks of exposure to TDF.
Time Frame: Baseline and 96 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 37 | 37 | 74
cells/mm^3 | -77 (408.3) | -56 (305.6) | -67 (358.3)

38. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 144 Weeks
Description: This is the change from baseline in CD4 cell count after 144 weeks of exposure to TDF.
Time Frame: Baseline and 144 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 33 | 38 | 71
cells/mm^3 | -139 (438.2) | -146 (245.3) | -142 (345.9)

39. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 192 Weeks
Description: This is the change from baseline in CD4 cell count after 192 weeks of exposure to TDF.
Time Frame: Baseline and 192 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 29 | 37 | 66
cells/mm^3 | -304 (529.0) | -177 (288.5) | -233 (413.2)

40. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 240 Weeks
Description: This is the change from baseline in CD4 cell count after 240 weeks of exposure to TDF.
Time Frame: Baseline and 240 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 27 | 32 | 59
cells/mm^3 | -369 (529.9) | -296 (252.6) | -329 (401.7)

41. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 288 Weeks
Description: This is the change from baseline in CD4 cell count after 288 weeks of exposure to TDF.
Time Frame: Baseline and 288 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 26 | 25 | 51
cells/mm^3 | -346 (507.5) | -256 (292.5) | -302 (414.6)

42. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 336 Weeks
Description: This is the change from baseline in CD4 cell count after 336 weeks of exposure to TDF.
Time Frame: Baseline and 336 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 23 | 22 | 45
cells/mm^3 | -415 (569.4) | -283 (252.2) | -350 (443.8)

43. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 384 Weeks
Description: This is the change from baseline in CD4 cell count after 384 weeks of exposure to TDF.
Time Frame: Baseline and 384 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 19 | 10 | 29
cells/mm^3 | -620 (635.6) | -305 (238.2) | -512 (548.8)

44. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 432 Weeks
Description: This is the change from baseline in CD4 cell count after 432 weeks of exposure to TDF.
Time Frame: Baseline and 432 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 14 | 7 | 21
cells/mm^3 | -795 (559.2) | -302 (355.2) | -631 (545.7)

45. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 480 Weeks
Description: This is the change from baseline in CD4 cell count after 480 weeks of exposure to TDF.
Time Frame: Baseline and 480 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 10 | 3 | 13
cells/mm^3 | -923 (755.4) | -448 (469.9) | -813 (712.9)

46. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at 528 Weeks
Description: This is the change from baseline in CD4 cell count after 528 weeks of exposure to TDF.
Time Frame: Baseline and 528 weeks
Population: Intent-to-treat, Missing = Excluded
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Tenofovir DF | (Stavudine or Zidovudine)/TDF | All TDF
Number analyzed (Participants) | 6 | 0 | 6
cells/mm^3 | -710 (447.0) |  | -710 (447.0)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported in the open-label randomized period (Weeks 0-48), and during the extension period when all participants received tenofovir DF.
Description: Tenofovir DF and Stavudine or Zidovudine groups: AEs were reported from baseline through last dose (up to Week 48) + 30 days. AEs with onset during the extension period were excluded.
  All TDF group: AEs were reported from baseline through last dose + 30 days (median duration of exposure = 330.7 weeks)
Arm/Group | Tenofovir DF | Stavudine or Zidovudine | All TDF
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49 | 0/89
Serious Adverse Events (participants affected / at risk) | 2/48 | 2/49 | 15/89
Other Adverse Events (participants affected / at risk) | 37/48 | 35/49 | 82/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=48) | Stavudine or Zidovudine (N=49) | All TDF (N=89)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Lymph node abscess (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Shigella infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=48) | Stavudine or Zidovudine (N=49) | All TDF (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 8
Dental caries (Gastrointestinal disorders) | 1 | 1 | 22
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 20
Gastritis (Gastrointestinal disorders) | 2 | 1 | 8
Vomiting (Gastrointestinal disorders) | 6 | 0 | 11
Pyrexia (General disorders) | 1 | 3 | 14
Abscess limb (Infections and infestations) | 1 | 1 | 5
Acarodermatitis (Infections and infestations) | 0 | 0 | 8
Bronchitis (Infections and infestations) | 2 | 1 | 6
Conjunctivitis (Infections and infestations) | 2 | 0 | 7
Fungal skin infection (Infections and infestations) | 0 | 0 | 6
Gastroenteritis (Infections and infestations) | 3 | 4 | 18
Impetigo (Infections and infestations) | 0 | 2 | 10
Lice infestation (Infections and infestations) | 0 | 1 | 5
Oral herpes (Infections and infestations) | 2 | 1 | 9
Otitis media (Infections and infestations) | 7 | 4 | 16
Pharyngitis (Infections and infestations) | 1 | 0 | 16
Pharyngotonsillitis (Infections and infestations) | 1 | 1 | 14
Sinusitis (Infections and infestations) | 3 | 1 | 5
Tinea versicolour (Infections and infestations) | 1 | 1 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 10
Varicella (Infections and infestations) | 0 | 1 | 10
Viral upper respiratory tract infection (Infections and infestations) | 17 | 17 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Headache (Nervous system disorders) | 1 | 0 | 14
Proteinuria (Renal and urinary disorders) | 1 | 1 | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 12
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years